CLINICAL TRIAL: NCT06223945
Title: Surgical and Anesthesiological-resuscitation Aspects of Therapeutic Tactics for Thrombotic and Hemorrhagic Complications in Patients With the New Coronavirus Infection COVID-19
Brief Title: Thrombohemorrhagic Complications of COVID-19
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Volgograd State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12/2024/01/12
Record Dates: First submitted 2024-01-22; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: COVID-19 (Coronavirus Disease 2019)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrombotic and hemorrhagic complications of COVID-19 (Active Comparator)
  Interventions: Diagnostic Test: Prevention algorithm
- Prevention of thrombohemorrhagic complications in COVID-19 (Active Comparator)
  Interventions: Diagnostic Test: Prevention algorithm

INTERVENTIONS:
Diagnostic Test: Prevention algorithm — Development of an algorithm for the prevention of thrombohemorrhagic complications

SUMMARY:
The nature of the planned study:

The topic is of an applied nature and is aimed at improving the results of comprehensive treatment of patients with COVID-19, the course of whose disease was complicated by thrombotic or hemorrhagic catastrophes.

It is planned to analyze the results of treatment of this category of patients based on the work of several centers that provided surgical care to patients with COVID-19 during the pandemic (8 cities).

As a result of the analysis, it is planned to develop algorithms for the prevention and treatment of thrombotic and hemorrhagic complications in patients with COVID-19.

The proposed study will be multicenter, cohort, retrospective.

The purpose of the study:

Improvement of treatment results in COVID-19 patients with thrombotic or hemorrhagic complications

Scientific novelty:

For the first time, as a result of a multicenter study, it is expected to identify the most effective approach to the treatment and prevention of thrombotic and hemorrhagic complications in patients with COVID-19.

For the first time, it is planned to develop and put into practice algorithms for the application of the most effective methods of treatment and prevention of thrombohemorrhagic complications of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thrombohemorrhagic complications who were treated in a covid hospital

Exclusion Criteria:

* Cancer patients
* Patients who had thrombohemorrhagic disorders before admission to the hospital
* Pregnant women
* Patients receiving routine anticoagulant and antiplatelet therapy before admission to the hospital

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2029-01-12 (Estimated); Study Completion 2029-01-12 (Estimated)

PRIMARY OUTCOMES:
development of an algorithm for the prevention of thrombohemorrhagic complications of COVID-19 | 5 years
  It is planned to perform a multicenter cohort retrospective study with an expanded analysis of the clinical features of the course, the results of surgical treatment, intensive care, anesthesiological and resuscitation benefits in patients with COVID-19, the course of which was complicated by thrombotic and hemorrhagic complications, including internal and external bleeding from the hollow organs of the abdominal cavity, retroperitoneal space and chest. The material for the study will be formed by combining data from several large clinics, on the basis of which infectious diseases hospitals with a concentration of surgical patients have been deployed. Based on the cumulative assessment of the results obtained, new and improved previously developed surgical and anesthetic-resuscitation algorithms for diagnosis, surgical tactics, intensive care in patients with COVID-19 with thrombotic and hemorrhagic complications in need of surgical and resuscitation procedures will be proposed.

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Mikhin, Study Chair — Volgograd State Medical University
Locations (1):
- Clinic №1 of Volgograd State Medical University, Volgograd, Russia